CLINICAL TRIAL: NCT00769912
Title: Evaluation of of a Prefixed 50% N2O- 50%O2 Mixture in Legal Abortion Under Local Analgesia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2008-000799-25; 2008-10
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2011-01

CONDITIONS: Abortion
MeSH Terms: interventions — Air

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 50% N2O- 50%O2 mixture administration during the intervention
  Interventions: Drug: 50% N2O- 50%O2 mixture
- 2 (Placebo Comparator): Placebo (air) during the intervention
  Interventions: Drug: Placebo (air)

INTERVENTIONS:
Drug: 50% N2O- 50%O2 mixture — 50% N2O- 50%O2 mixture administration
  Arms: 1
Drug: Placebo (air) — Placebo administration during the intervention
  Arms: 2

SUMMARY:
To evaluate effectiveness of a prefixed 50% N2O- 50%O2 mixture in legal abortion under paracervical block.

ELIGIBILITY:
Inclusion Criteria:

* Major patient having signed an assent waits having chosen to make the intervention under local anesthetic

Exclusion Criteria:

* Minor
* contraindication in the use of the paracetamol, the lidocaine
* Porphyries

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2008-10; Primary Completion 2009-02 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Pain during the intervention | 4 months

SECONDARY OUTCOMES:
Pain at the end of the intervention and 2 hours after. Unwanted events | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Aubert AGOSTINI, MD, Principal Investigator — Assistance Publique des Hopitaux de Marseille
Locations (1):
- Service de Gynécologie Obstétrique, Hôpital La Conception, Marseille, France